CLINICAL TRIAL: NCT06459856
Title: Combined Effects of Balloon Blowing Therapy With Percussion on Pulmonary Functions in Patients With Pneumonia
Brief Title: Combined Effects of Balloon Blowing Therapy With Percussion in Patients With Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0371
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia
Keywords: Balloon Therapy, Percussion, Pneumonia, Breath Sounds
MeSH Terms: conditions — Pneumonia; Respiratory Sounds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon Blowing, Percussion (Experimental): intervention will be given as blowing 10-15 balloons per day for 6 days. 05.minutes active cycle of breathing technique as baseline 10 minute to blowing 15 balloons 10 minutes percussion 25 minutes session
  Interventions: Other: Balloon blowing; Other: Percussion
- Perccussion (Active Comparator): intervention Will be given as Buteyko breathing techniques for 3 weeks. 15 Minutes ACBT with rest interval 10 minutes percussion 25 minutes session
  Interventions: Other: Percussion

INTERVENTIONS:
Other: Balloon blowing — Ask the patient to take in a deep breath; steadily and slowly blow up the huge balloon. See the balloon getting bigger, and bigger. Now ask the patient to close the eyes and imagine the balloon floating into the air. Let the patient continue blowing of balloons until he or she gets relaxed and calm.
  Arms: Balloon Blowing, Percussion
Other: Percussion — Percussion is a technique involving rhythmic tapping or clapping on the chest or back, serves as a means to move and loosen retained secretions within the airways. This mechanical intervention helps in removing mucus from the bronchial walls, and facilitates its expectoration and clearance

SUMMARY:
Pneumonia is an infection of the lungs that is caused by bacteria, viruses, fungi, or parasites. It is characterized primarily by inflammation of the alveoli in the lungs or by alveoli that are filled with fluid (alveoli are microscopic sacs in the lungs that absorb oxygen). The symptoms of pneumonia can develop suddenly (over 24-48 hours) or may show more slowly, over several days. Common symptoms of pneumonia are likely to have a cough which can be dry, or may produce phlegm (thick mucus) that is yellow, green, brownish or bloodstained and breathing difficulty, wheezing and chest tightness where the rate will be high and the rhythm will be rapid and shallow. This activity encourages deep breathing, allowing a patient body to relax. Explain the patient that this exercise will help him or he can feel more relaxed. Make the patient to imagine that he/she is blowing up a balloon. Ask him/her to take in a deep breath; steadily and slowly blow up the huge balloon. See the balloon getting bigger, and bigger. Now ask the patient to close the eyes and imagine the balloon floating into the air. Let the patient continue blowing of balloons until he or she gets relaxed and calm. Percussion is a technique involving rhythmic tapping or clapping on the chest or back, serves as a means to move and loosen retained secretions within the airways. This mechanical intervention helps in removing mucus from the bronchial walls, and facilitates its expectoration and clearance.

DETAILED DESCRIPTION:
Pneumonia is an infection of the lungs that is caused by bacteria, viruses, fungi, or parasites. It is characterized primarily by inflammation of the alveoli in the lungs or by alveoli that are filled with fluid (alveoli are microscopic sacs in the lungs that absorb oxygen). The symptoms of pneumonia can develop suddenly (over 24-48 hours) or may show more slowly, over several days. Common symptoms of pneumonia are likely to have a cough which can be dry, or may produce phlegm (thick mucus) that is yellow, green, brownish or bloodstained and breathing difficulty, wheezing and chest tightness where the rate will be high and the rhythm will be rapid and shallow. This activity encourages deep breathing, allowing a patient body to relax. Explain the patient that this exercise will help him or he can feel more relaxed. Make the patient to imagine that he/she is blowing up a balloon. Ask him/her to take in a deep breath; steadily and slowly blow up the huge balloon. See the balloon getting bigger, and bigger. Now ask the patient to close the eyes and imagine the balloon floating into the air. Let the patient continue blowing of balloons until he or she gets relaxed and calm. Percussion is a technique involving rhythmic tapping or clapping on the chest or back, serves as a means to move and loosen retained secretions within the airways. This mechanical intervention helps in removing mucus from the bronchial walls, and facilitates its expectoration and clearance.

This research methodology is likely to employ a randomized clinical trial design, dividing participants into two groups: group A will be receiving the combined therapy (Balloon blowing, percussion) for 7 days, while the Group B will be given intervention as Buteyko breathing techniques (ACBT, Percussion and deep breathing) for 3 weeks. Parameters such as breath auscultation by stethoscope, CASA Q questionnaire, Pulmonary function test will likely be utilized to gauge the efficacy of the combined intervention versus standard treatments. Anticipated outcomes encompass improvements in lung function metrics, clearer breath sounds denoting improved airway clearance, and potentially quicker recovery or shortened illness duration as compared to conventional treatments. If successful, this study could signify a more comprehensive and effective approach to manage pneumonia by combining specific therapies to enhance pulmonary functions and help in patients' recovery. Ultimately, these findings could contribute significantly to use respiratory therapy for individuals suffering from pneumonia

ELIGIBILITY:
Inclusion Criteria:

• Diagnosed pneumonia patients

Exclusion Criteria:

* Other respiratory complications
* Patients with surgeries
* Patients with neurological disorders

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
FEV1(Forced Expiratory Volume per second) | Pre and post after 1 week
  Pulmonary Function Test using Digital Spirometer
FVC (Forced Vital Capacity) | Pre and Post after 1 week
  Pulmonary Function Test using Digital Spirometer
FEV1/FVC | Pre and Post after 1 week
  Pulmonary Function Test using Digital Spirometer
CASA-Q (Cough and Sputum Assessment Questionnaire) | Pre and post after 1 week
  To assess the Level of Cough and Sputum
Auscultatory Breath Sound | pre and Post after 1 week
  To assess the breath sound

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Shehzadi, Mphil, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore Teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No